CLINICAL TRIAL: NCT06780995
Title: Power Exercise for Stroke Recovery: A Pilot Randomized Controlled Trial (POWER-Pilot)
Brief Title: Power Exercise for Stroke Recovery: The POWER Pilot Trial (POWER-P)
Acronym: POWER-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ada Tang, Professor, Assistant Dean, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: POWER-Pilot
Record Dates: First submitted 2024-12-09; First posted 2025-01-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Stroke; Aging; Resistance training; Power training; Physical function; Community exercise; Quality of life; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power Exercise for Stroke Recovery (POWER) (Experimental): POWER involves 3 progressive phases: 1) Familiarization (1 week), 2) Strength (4 weeks, 2-3 sets, 5-8 repetitions), and 3) Power (5 weeks, 2-3 sets, 15-20 repetitions, fast tempo).
  Interventions: Other: Power Exercise for Stroke Recovery (POWER)
- Strength Training Engaging Guidelines to Enhance Total Health (STRENGTH) (Active Comparator): STRENGTH is based on current resistance exercise training (RET) clinical practice guidelines for stroke with no focus on power.
  Interventions: Other: Strength Training Engaging Guidelines to Enhance Total Health (STRENGTH)

INTERVENTIONS:
Other: Power Exercise for Stroke Recovery (POWER) — POWER incorporates 3 progressive phases: Phase 1 Familiarization (Week 1) as a low-intensity version of the training program to acclimate participants to the movements (body weight resisted or light weights, RPE 2-3 "Fairly light" to "Moderate"). Phase 2 Strength (Weeks 2-5) progresses loads to achieve volitional fatigue within 6-8 repetitions (RPE 7-9 "Very hard" to "Very very hard"). Phase 3 Power (Weeks 6-10) will use intensities RPE 4-6 ("Somewhat hard" to "Very hard"), and exercises will be executed at the highest possible velocity to focus on muscle power. The Power phase is intentionally designed with exercises to emphasize functional movements such as fast sit to stands, lunging and calf raises.
  Arms: Power Exercise for Stroke Recovery (POWER)
Other: Strength Training Engaging Guidelines to Enhance Total Health (STRENGTH) — STRENGTH is based on current clinical practice guidelines for RET after stroke. It will include the same Familiarization week as the POWER program (Week 1), followed by progressive conventional RET involving 3 sets of 10-15 repetitions at moderate to high intensities (RPE 4-5 "Somewhat hard" to "Hard") (Weeks 2-10). The external resistance will be progressed to maintain this target RPE range. STRENGTH is matched with POWER in length (60-minute sessions over 10 weeks), frequency (3x/week) and format (in-person supervision).
  Arms: Strength Training Engaging Guidelines to Enhance Total Health (STRENGTH)

SUMMARY:
Weakness is one of the most common consequences of stroke. For the over 750,000 Canadians living with stroke, many daily activities like standing from a chair, walking and balance not only require strength but often efforts in bursts, known as muscle power. Strength training can improve muscle strength and, when performed at higher speeds, can help build muscle power. Current guidelines for stroke recommend strength training but these are commonly performed at lower intensities and do not include any focus on building muscle power. There has been very little research on power training after stroke.

A 10-week power training program for people living with stroke, Power Exercise for Stroke Recovery (POWER-Feasibility, NCT05816811) was recently evaluated. POWER includes 3 phases of progressive exercise: building familiarity with the upper and lower body exercises, then strength, and lastly muscle power. The results from POWER-Feasibility are promising, suggesting that POWER is safe and may improve stroke recovery. POWER-Feasibility was a small study (15 participants), and POWER was not compared to a control intervention.

A pilot randomized controlled trial of POWER (POWER-Pilot) will now be conducted. Sixty people who are at least 6 months after stroke will be recruited. They will be randomly assigned to participate in POWER or standard strength training for stroke at lower intensities and without focus on power training. The feasibility of a randomized study will be examined, and whether POWER can improve walking, strength and balance compared to the control group. Results from POWER-Pilot will help design a larger randomized trial in the future (POWER-RCT), and may ultimately be important for stroke rehabilitation teams to better understand whether power training can help people recovering from stroke.

DETAILED DESCRIPTION:
With the population aging, nearly 750,000 Canadians live with stroke, surpassing previous projections by 15 years. Post-stroke deficits, including loss of strength, balance and walking ability, are highly common. Sarcopenia, often associated with aging yet highly prevalent in stroke, underlie these deficits and contribute to lower discharge rates after hospitalization.

Community stroke exercise programs can improve strength and function to aid in recovery beyond hospital care. Most programs however follow conservative resistance exercise training (RET) approaches, as stroke guidelines are based on limited evidence. Unlike benefits of RET shown in mobility in older adults, stroke trials have shown large improvements in strength without concurrent changes in mobility, motor function or walking.

Power-focused RET involves moving lighter weights at high speed to develop muscle power, which may be more important than strength alone for activities critical for independent living such as climbing stairs, balance, and walking speed. A novel, progressive power training-focused community program for stroke (Power Exercise for Stroke Recovery, POWER) was developed to influence recovery of physical function. Following a successful single-group feasibility study of POWER (POWER-Feasibility, NCT05816811), a phase II pilot randomized trial (POWER-Pilot) is needed.

This pilot randomized trial aims to answer the following questions: 1) What is the feasibility of a multi-site randomized design to evaluate Power Exercise for Stroke Recovery (POWER), a power-focused training program for people living in the community with stroke? 2) What are the preliminary estimates of the effect of POWER compared to conventionally recommended RET (Strength Training Engaging Guidelines to Enhance Total Health, STRENGTH) for people living in the community with stroke on outcomes of functional mobility (walking, balance), post-stroke fatigue, psychological wellbeing, cognition, and health-related quality of life?

Sixty participants (6 months post-stroke, completed rehabilitation) will be randomized to POWER or STRENGTH. POWER involves 3 progressive phases: 1) Familiarization (1 week), 2) Strength (4 weeks, 2-3 sets, 5-8 repetitions), and 3) Power (5 weeks, 2-3 sets, 15-20 repetitions, fast tempo). STRENGTH is based on current RET clinical practice guidelines for stroke with no focus on power. POWER and STRENGTH matched in length, frequency (3x/week) and format (in-person supervision) but differentiated by approach to exercise progression, intensity, and tempo.

Feasibility indicators such as randomization and blinding have predefined success and progression thresholds. Estimates of the effect of POWER include functional mobility (Timed Up and Go, primary clinical outcome), walking speed, post-stroke fatigue, psychological well-being, cognition, balance, and quality of life, and will be assessed pre-post, and at 8-week follow-up. Sex and gender-related factors associated with feasibility and changes in clinical outcomes as social determinants of exercise participation post-stroke will also be examined.

Feasibility outcomes and effect estimates from POWER-Pilot will guide scalability for a fully powered RCT and future cost-effectiveness evaluation, shaping exercise best practices and facilitating hospital-to-community transition through broader implementation in community programs.

ELIGIBILITY:
Inclusion Criteria:

1. ≥19 years old
2. ≥6 months poststroke,
3. able to walk >10 meters with or without an assistive device
4. have mild to moderate stroke severity (modified Rankin Scale ≤3)
5. without significant cognitive impairment that would preclude safe exercise, screened via Montreal Cognitive Assessment-Blind score <18

Exclusion Criteria:

1. Any contraindications to exercise for people with cardiovascular disease, such as unstable angina, uncontrolled hypertension, orthostatic blood pressure with exercise, or uncontrolled arrhythmias or
2. Actively engaged in or have made plans to engage in stroke rehabilitation services

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Randomization - Percentage of participants allocated as assigned | Through study completion, over 24 months
  Indicator: Yes/No; Criteria for success and progression: Success: 100% participants allocated as assigned, Revise: <100% participants allocated as assigned
Feasibility: Randomization - Clinically important difference between groups | Through study completion, over 24 months
  Indicator: Balance of prognosis; Criteria for success and progression: Success: No clinically important differences between groups, Revise: Clinically important differences between groups
Feasibility: Allocation concealment | Through study completion, over 24 months
  Indicator: Yes/No; Criteria for success and progression: Success: Allocation concealment preserved, Revise: Allocation revealed
Feasibility: Assessor blinding - Number of occurrences of unblinding | Through study completion, over 24 months
  Indicator: # occurrences of unblinding; Criteria for success and progression: Success: Assessors unblinded for <5% of participants, Revise: Assessors unblinded for ≥5% of participants
Feasibility: Contamination - Number of participants exposed to other intervention arm | Through study completion, over 24 months
  Indicator: # participants exposed to the other intervention arm; Criteria for success and progression: Success: No occurrences of contamination, Revise: Any occurrence of contamination
Feasibility: Recruitment rate - Number of participants recruited per month | Through study completion, over 24 months
  Indicator: # recruited / month; Criteria for success and progression: Success: Mean 1.0 participants/month/site, Revise: Mean <1.0 participants/month/site
Feasibility: Retention rate - Percentage of participants with follow up data | Through study completion, over 24 months
  Indicator: % follow up data; Criteria for success and progression: Success: Complete follow up data in ≥80% participants, Revise: Complete follow up data in <80% participants
Feasibility: Participant and assessor burden - Percentage of participants completing study assessments in ≤1.5h | Through study completion, over 24 months
  Indicator: time to complete assessments; Criteria for success and progression: Success: ≥80% complete assessments in ≤1.5h, Revise: <80% complete assessments in ≤1.5h
Feasibility: Participant and assessor burden - Participant rating of the burden of assessments | Through study completion, over 24 months
  Indicator: perceived burden of assessments; Criteria for success and progression: Success: Rating ≤3 on 10-point Likert scale (1=not at all; 10=extremely burdensome), Revise: Rating >3 out of 10
Feasibility: Safety - Number of serious adverse events | Through study completion, over 24 months
  Indicator: Serious adverse events from assessments or interventions; Criteria for success and progression: Success: 0 occurrences, Revise: Any occurrences
Feasibility: Treatment effect - Availability of clinical outcome data | Through study completion, over 24 months
  Indicator: Number of available data points at post-intervention; Criteria for success and progression: ≥90% (n=54/60) data available on all clinical outcomes of interest
Functional mobility: Timed Up and Go (TUG) test (self- and fast-paced) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Timed Up and Go is a measure of functional mobility. A standard chair (~46cm in height) will be placed at the start of a flat walking course and a cone will be placed 3 meters from the chair. Participants will stand from the chair, walk 3 meters, turn back towards the chair, and sit back down, without assistance. This will be completed at a comfortable pace and fast pace. The task will be timed and measured in seconds, a shorter time indicates better mobility and balance.

SECONDARY OUTCOMES:
Walking speed: 10-meter walking speed (self- and fast-paced) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  Participants will be instructed to walk a total of 14 meters, including 2-meter initiation and termination phases. Their walking pace was assessed across the 10-meter distance between these two points. The middle ten meters of a fourteen-meter walkway will be timed. This will be completed at the participant's comfortable walking pace and at their fast pace. The average of two trials will be determined for each pace.
Post-stroke fatigue: Fatigue Severity Scale-7 (FFS) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Fatigue Severity Scale is a 9-item questionnaire that uses a 7-point Likert scale to measure fatigue and its impact on an individual's activities and lifestyle: The scale ranges from 1, which means "strongly disagree", to 7, which means "strongly agree". The minimum score is 9, and the maximum is 63 with higher scores indicating greater fatigue severity.
Psychological well-being: General Health Questionnaire-28 | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  General Health Questionnaire-28 assesses ability to carry out daily functions and appearances of new signs and symptoms across 4 domains (somatic symptoms, anxiety/insomnia, social function, severe depression). It uses a Likert scale with "Not at all" scored as 0, "No more than usual" as 1, "Rather more than usual" as 2, and "Much more than usual" as 3. The total score ranges from 0 to 84, with higher scores indicating greater psychological distress. Subscale scores are calculated by summing the scores of the seven items within each of the four subscales.
Cognition: Montreal Cognitive Assessment (MoCA) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Montreal Cognitive Assessment is a brief screening test for detecting mild cognitive impairments. It assesses executive functioning, visuospatial abilities, memory, attention, working memory, language, and orientation. It is scored out of a total of 30 points, with higher scores indicating better cognitive function.
Standing balance: Brief Balance Evaluation System Test (Brief BESTest) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Brief BESTest consists of 6 items that assess 6 different aspects contributing to postural control in standing and walking. It is scored based on a series of 14 items that assess balance in individuals, with each item scored on a 0 to 3 scale, where 0 indicates the lowest level of balance function and 3 indicates the highest. The total score is calculated by summing the individual item scores, with a possible range of 0 to 42. Higher scores reflect better balance performance.
Standing balance: Berg Balance Scale (BBS) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Berg Balance Scale is scored based on 14 items that assess various aspects of balance, such as sitting, standing, reaching, and turning. Each item is rated on a 5-point scale, where 0 indicates the lowest level of function and 4 indicates the highest. The total score is obtained by summing the individual scores, with a possible range of 0 to 56. A higher score indicates better balance and lower risk of falls.
Health-related quality of life: Stroke Impact Scale 3.0 (SIS 3.0) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Stroke Impact Scale 3.0 is scored based on 59 items across 8 domains, including strength, memory, emotion, hand function, mobility, communication, activities of daily living, and participation. Respondents rate their experiences or abilities in each domain on a 5-point Likert scale, with higher scores indicating better function or less impairment. The individual domain scores are transformed into a scale ranging from 0 to 100, with 100 representing the best possible outcome.
Health-related quality of life: EuroQol-5D-5L (EQ-5D-5L) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The EuroQol-5D-5L is a brief, generic, health status measure composed of 5 questions with Likert response options (descriptive system) and a visual analog scale (EQ-VAS). Each dimension has five levels of severity, ranging from no problems (level 1) to extreme problems (level 5). The scores for each dimension are combined to create a health state profile, which can be transformed into a single summary index score ranging from 0 to 1, with higher scores representing better health.
Participation: Measure of Experiential Aspects of Participation (MeEAP) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Measure of Experiential Aspects of Participation is a measure to evaluate the quality of participation for people with disabilities across employment, mobility, and sport and exercise life domains. The scoring involves assigning numerical values to each item based on the frequency, satisfaction, and importance of the activities, with higher scores indicating greater perceived quality and value of participation.
Lower extremity strength and endurance: 30-second chair stand test (30sCST) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The 30-second chair stand test is a measure of lower extremity strength and endurance. It is scored based on the number of times an individual can rise from a seated position to a full standing position and sit back down within 30 seconds.The score is determined by counting the total number of complete stands performed within the 30-second time limit. A higher score indicates better lower body strength and endurance.
Self-efficacy for balance: Activities-Specific Balance Confidence Scale (ABC) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Activities-Specific Balance Confidence Scale is a structured questionnaire that measures an individual's confidence during ambulatory activities. It is scored based on a participant's confidence in performing 16 daily activities without losing balance or becoming unsteady. Each item is rated on a scale from 0 to 100, where 0 indicates no confidence and 100 indicates complete confidence. The scores for all 16 items are averaged to produce an overall score, with higher scores reflecting greater confidence in balance during everyday activities.
Confidence in exercising: Exercise Self-Efficacy Scale (ESES) | Baseline (0 weeks), post-intervention (10 weeks), follow-up (18 weeks)
  The Exercise Self-Efficacy Scale is a patient reported outcome measure consisting of 10 items, which assess confidence in exercising under certain circumstances. Participants rate their confidence on a 4-point scale ranging from 1 (Not always true) to 4 (Always true).
Responsiveness to outcome measures: Global Rating of Change (GRC) questionnaire | Post-intervention (10 weeks)
  The Global Rating of Change questionnaire will be used to examine the responsiveness of the outcome measures. Participants are asked: "With respect to the following areas, how would you describe yourself now compared to when you started the study?" Participants will rate their change on a scale ranging from 1 to 5, where 1 indicated much worse and 5 indicated much better compared to the start of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The University of British Columbia - Okanagan Campus, Kelowna, British Columbia
  - McMaster University, Hamilton, Ontario